CLINICAL TRIAL: NCT02736747
Title: Immediate Effects of Cryotherapy on Neuromuscular Performance of Ankle Joint and on Gait Pattern of Chronic Spastic Hemiparetic Subjects Post-Stroke
Brief Title: Effects of Cryotherapy on Ankle Movements and Gait of Spastic Hemiparetic Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Carolina Carmona de Alcântara (Other)
Responsible Party: Sponsor-Investigator, Carolina Carmona de Alcântara, PhD student, Universidade Federal de Sao Carlos
Organization: Universidade Federal de Sao Carlos (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Cryotherapy_LAFIN
Record Dates: First submitted 2016-03-18; First posted 2016-04-13 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Stroke; Muscle Spasticity
Keywords: Stroke; Muscle Spasticity; Cryotherapy; Gait; Muscle Weakness; Proprioception
MeSH Terms: conditions — Stroke; Muscle Spasticity; Muscle Weakness | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cryotherapy (ice pack) (Active Comparator): A pack with 1000g of crushed ice without air will be placed for 20 consecutive minutes on a pre-delimited rectangular area with dimensions of 25 x 35 cm and will be fixed with a non-compressive elastic band. One strip of plastic paper will encompass the paretic leg of the subjects, avoiding direct contact from the skin with the ice pack.
  Interventions: Other: Cryotherapy
- Placebo (sand pack) (Placebo Comparator): For placebo application, the pack will be filled with 1000g of thin sand, in environmental temperature, so that the pressure exerted will be the same as the ice pack. All other experimental procedures will follow the same protocol as "cryotherapy application".
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Cryotherapy
  Arms: Cryotherapy (ice pack)
Other: Placebo
  Arms: Placebo (sand pack)

SUMMARY:
The stroke has been described as the third cause of death and main cause of disability in the worldwide population. About 60% of the survivors are able to walk following the rehabilitation process, however deficits on lower limbs functions often persists in most cases, affecting the gait and functional mobility. In this sense, several interventions are applied in the clinical practice to optimize the functional performance. Cryotherapy is one of the most used techniques aiming to reduce spasticity temporarily, allowing the training of functional tasks, such as walking. The aim of the present study is to evaluate the immediate effects of cryotherapy (ice pack) on neuromuscular performance, proprioception, passive resistance of dorsiflexors and plantarflexors muscles, and also on gait performance in chronic post-stroke subjects. Eighteen chronic hemiparetic subjects will participate in this crossover placebo-controlled trial. The order of intervention (cryotherapy or placebo) will be randomized. Fifteen days of washout period will be considered. The cryotherapy/placebo will be applied on the posterior area of the leg for 20 minutes. Initially Fugl Meyer will be applied. All other assessments will be performed before and after intervention: spasticity level, classified according to Modified Ashworth Scale; temporo-spatial and angular parameters for trunk, hip, knee and ankle during gait, using a motion analysis system (Qualysis AB, Gothenburg, Sweden); the proprioception (joint position sense), passive resistance to stretching, isometric and isokinetic torques during contractions of plantarflexors and dorsiflexors of the ankle, evaluated through isokinetic dynamometer. Concomitantly, bilateral activation of soleus, gastrocnemius, tibialis anterior and peroneus will be assessed by electromyography during isokinetic dynamometer assessment and gait. The following electromyographic variables will be analyzed: maximum activation amplitude, muscle onset, coactivation index between agonists and antagonists. For statistical analysis, normality (Shapiro Wilk) and homogeneity (Levene) tests will be applied. If the variables have a distribution considered normal and homogeneous, Two-way ANOVA with repeated measures will be applied. Otherwise, non-parametric statistics (Friedman test) will be applied. A significance level of 0.05 will be considered for all statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke (last episode of stroke occurred more than 6 months ago)
* Ischemic stroke
* Minimum score on the Mini Mental State Examination, according to the subject's educational level
* Spasticity level between 1 and 4 according to Modified Ashworth Scale for the plantarflexors
* Locomotion capacity of 2 to 4 according to Functional Ambulation Category (FAC).

Exclusion Criteria:

* Diabetic peripheral neuropathy
* Adverse reactions to cold
* Intolerance to cold application
* Absence of sensibility to cold
* Diagnostic of Raynaud syndrome
* Ulcers or skin lesions
* Severe cardiovascular or peripheral vascular diseases (heart failure, arrhythmias, angina pectoris, and acute myocardial infarction)
* Other neurological or orthopedic diseases
* Toxin bothulinium injection 4 months or sooner
* Cognitive impairments
* Any history of joint or muscle injuries of the lower limbs
* Body mass index (BMI) greater than 28 kg/m²
* Pain during the any experimental procedure.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-04; Primary Completion 2017-07 (Actual); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in spasticity level | baseline, 20 minutes (immediately post-application of cryotherapy or placebo)
  Spasticity level of plantarflexors and dorsiflexors will be classified according to Modified Ashworth Scale.
Change from baseline in angular kinematic variables during gait | baseline, 20 minutes (immediately post-application of cryotherapy or placebo)
  The post-evaluation will be performed immediately after the end of the intervention (cryotherapy or placebo, applied for 20 minutes). A motion analysis system (Qualysis AB, Gothenburg, Sweden) will be used for kinematic data collection during gait. Passive reflective markers will be placed on the anatomical landmarks (anatomical markers) according to the International Society of Biomechanics. In addition, clusters will be placed on T4, L2 and bilaterally on the lateral portion of the thighs and legs. Following markers and clusters placement, a static posture (duration: 10 seconds) will be performed with the subjects in orthostatic position. Then dynamic data will be collected during walking in the self-selected comfortable speed (10 trials). The displacement (°) of the joints of the trunk, hip, knee and ankle during heel strike, stance phase and balance phase will be calculated during gait.
Change from baseline in linear kinematic variables during gait | baseline, 20 minutes (immediately post-application of cryotherapy or placebo)
  The post-evaluation will be performed immediately after the end of the intervention (cryotherapy or placebo, applied for 20 minutes). A motion analysis system (Qualysis AB, Gothenburg, Sweden) will be used for kinematic data collection during gait. Passive reflective markers will be placed on the anatomical landmarks (anatomical markers) according to the International Society of Biomechanics. In addition, clusters will be placed on T4, L2 and bilaterally on the lateral portion of the thighs and legs. Following markers and clusters placement, a static posture (duration: 10 seconds) will be performed with the subjects in orthostatic position. Then dynamic data will be collected during walking in the self-selected comfortable speed (10 trials) and linear kinematic variables during gait will be analyzed.
Change from baseline in joint sense position (proprioception) during plantarflexion and dorsiflexion | baseline, 20 minutes (immediately post-application of cryotherapy or placebo)
  The post-evaluation will be performed immediately after the end of the intervention (cryotherapy or placebo, applied for 20 minutes). The joint position sense (proprioception) test will be performed on an isokinetic dynamometer. The participants will be seated and blindfolded. Initially, the dynamometer will move the foot toward references angles (for dorsiflexion or plantarflexion). Then, subjects will be allowed to sense the reference angle for 10 seconds before the ankle is returned passively to the start position. Subsequently, the foot will be moved passively by the dynamometer toward the reference position (for dorsiflexion or plantarflexion), and subjects will press a button in their hand that will stop the machine when they feel the position has been reached. The absolute error (in degrees) will be calculated as the difference between the indicated and reference positions.
Change from baseline in passive resistance of plantarflexors and dorsiflexors | baseline, 20 minutes (immediately post-application of cryotherapy or placebo)
  The post-evaluation will be performed immediately after the end of the intervention (cryotherapy or placebo, applied for 20 minutes). The assessment of passive resistance for plantarflexion and dorsiflexion muscles will be performed on an isokinetic dynamometer. The equipment will passively move the foot in a series of 6 repetitions in the movements of dorsiflexion and plantar flexion. Both responses to slow and fast passive stretching will be evaluated. Passive torque peak (N.m) of plantarflexors and dorsiflexors of the ankle will be recorded.
Change from baseline in torque during isometric contractions | baseline, 20 minutes (immediately post-application of cryotherapy or placebo)
  The post-evaluation will be performed immediately after the end of the intervention (cryotherapy or placebo, applied for 20 minutes). The isometric active torques (N.m) generated during plantarflexion and dorsiflexion contractions will be assessed using an isokinetic dynamometer.
Change from baseline in torque during concentric contractions | baseline, 20 minutes (immediately post-application of cryotherapy or placebo)
  The post-evaluation will be performed immediately after the end of the intervention (cryotherapy or placebo, applied for 20 minutes). The active torques generated (N.m) during plantarflexion and dorsiflexion movements will be assessed using an isokinetic dynamometer.
Change from baseline in torque during eccentric contractions | baseline, 20 minutes (immediately post-application of cryotherapy or placebo)
  The post-evaluation will be performed immediately after the end of the intervention (cryotherapy or placebo, applied for 20 minutes). The active torques generated (N.m) during plantarflexion and dorsiflexion movements will be assessed using an isokinetic dynamometer.
Change from baseline in electromyography assessment | baseline, 20 minutes (immediately post-application of cryotherapy or placebo)
  The post-evaluation will be performed immediately after the end of the intervention (cryotherapy or placebo, applied for 20 minutes). Bilateral activation of soleus, gastrocnemius, tibialis anterior and peroneus will be assessed by electromyography concomitantly with isokinetic dynamometer and gait assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Thiago L. Russo, PhD, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Universidade Federal de São Carlos, São Carlos, São Paulo, Brazil

REFERENCES:
- [Derived] Alcantara CC, Blanco J, De Oliveira LM, Ribeiro PFS, Herrera E, Nakagawa TH, Reisman DS, Michaelsen SM, Garcia LC, Russo TL. Cryotherapy reduces muscle hypertonia, but does not affect lower limb strength or gait kinematics post-stroke: a randomized controlled crossover study. Top Stroke Rehabil. 2019 May;26(4):267-280. doi: 10.1080/10749357.2019.1593613. PMID 31012824